CLINICAL TRIAL: NCT01017848
Title: Urine pH as a Predictor of Diabetes
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, Associate Chair of Medicine, Northwell Health
Other Study IDs: 09-031
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes
Keywords: diabetes; urine pH; insulin resistance; metabolic syndrome; development of diabetes
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adults, nondiabetics: adults who are nondiabetic, no CKD, no urinary tract infection, no bladder dysfunction

SUMMARY:
Urine pH has been lately linked to insulin resistance. The early phase of Diabetes Mellitus involves insulin resistance. Thus, the investigators want to check if a simple cheap study like a urine analysis that can predict diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age > 18

Exclusion Criteria:

* diabetes
* CKD
* urine infection
* UTO
* bladder dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult inpatients, nondiabetic, no CKD, no urine infection, no UTO
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
development of diabetes using a predicting formula | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne El-Sayegh, MD, Principal Investigator — SIUH
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States